CLINICAL TRIAL: NCT04879316
Title: Analysis of Nutritional Biomarkers to Predict the Efficacy of Immunotherapy by Anti-PD/PDL1 Checkpoints Inhibitors in Metastatic Non-small Cell Lung Cancer Patients
Brief Title: Energy for Lymphocytes
Acronym: ELY
Status: Completed | Type: Observational
Sponsor: Hôpital Cochin (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Camille Levalois, Co-investigator, Hôpital Cochin
Other Study IDs: HCochin
Record Dates: First submitted 2021-04-12; First posted 2021-05-10 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Non-small Cell Lung Cancer; Progression, Disease
Keywords: cachexia; immunotherapy; carcinoma; Non-small cell lung cancer; Basal metabolism; Energy expenditure; inflammation; 6-month Progression free survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease Progression; Cachexia; Carcinoma; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult patients with NSCLC initiating nivolumab or pembrolizumab: Patients underwent a multidisciplinary evaluation including consultation with an oncologist and a dietitian. Such an assessment includes subjective and objective parameters such as medical history, weight loss, current dietary intake (including energy and protein balance), physical examination and anthropometric measurements, functional and mental assessment, medications, Resting Energy Expenditure measurement using indirect calorimetry and laboratory values.
  Interventions: Other: Resting Energy Expenditure measurement

INTERVENTIONS:
Other: Resting Energy Expenditure measurement — Resting Energy Expenditure measurement using indirect calorimetry

SUMMARY:
CERTIM is a cohort created in July 2015 to set up a multidisciplinary follow-up of cancer patients treated with immune checkpoint inhibitors.

From the CERTIM cohort, we conducted a longitudinal, prospective, observational study (ELY) in two tertiary university centers (Cochin hospital and European Georges Pompidou Hospital), which included patients between August 2016 and October 2019 and ended follow-up in April 2020.

Patients were treated with nivolumab, at a dose of 3 mg/kg every 2 weeks, or pembrolizumab, at a dose of 2mg/kg every 3 weeks. The investigators report findings from an evaluation of rest energy expenditure (REE) assessed using indirect calorimetry in the outpatient setting before treatment with checkpoints inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Stage IV histologically proven Non Small Cell Lung Cancer (NSCLC)
* Monotherapy with nivolumab or pembrolizumab.
* Patients were required to have measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.

Exclusion Criteria:

* Active malignancy other than NSCLC,
* ALK or EGFR mutated NSCLC
* Anticancer therapy or surgery within the past 2 weeks or inability to breathe under the calorimetry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with NSCLC initiating nivolumab or pembrolizumab in real-life conditions
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
6-month Progression-free survival | 6 months after start of treatment
  Calculated as the percentage of participants alive and without disease progression, as assessed by the Investigator using RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Derived] Montegut L, Joseph A, Chen H, Abdellatif M, Ruckenstuhl C, Motino O, Lambertucci F, Anagnostopoulos G, Lachkar S, Dichtinger S, Maiuri MC, Goldwasser F, Blanchet B, Fumeron F, Martins I, Madeo F, Kroemer G. High plasma concentrations of acyl-coenzyme A binding protein (ACBP) predispose to cardiovascular disease: Evidence for a phylogenetically conserved proaging function of ACBP. Aging Cell. 2023 Jan;22(1):e13751. doi: 10.1111/acel.13751. Epub 2022 Dec 12. PMID 36510662